CLINICAL TRIAL: NCT04004702
Title: Levetiracetam for Alzheimer's Disease Neuropsychiatric Symptoms Related to Epilepsy Trial (LAPSE) - A Phase II Exploratory Study
Brief Title: Levetiracetam for Alzheimer's Disease Neuropsychiatric Symptoms Related to Epilepsy Trial (LAPSE)
Acronym: LAPSE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06272019
Record Dates: First submitted 2019-06-27; First posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Alzheimer Disease
Keywords: neuro-psychiatric symptoms
MeSH Terms: conditions — Alzheimer Disease | interventions — Levetiracetam

STUDY DESIGN:
Intervention Model Description: Participants with clinical Alzheimer's disease and neuro-psychiatric symptoms will all be assessed with electroencephalogram, and all participants with epileptiform discharges will receive levetiracetam. Those without epileptiform discharges will be followed with serial inventories of symptom severity and functioning, but will not receive experimental treatment nor placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Levetiracetam (Experimental): All patients with epileptiform activity on initial screening EEG will receive levetiracetam for 1 year
  Interventions: Drug: Levetiracetam

INTERVENTIONS:
Drug: Levetiracetam — Levetiracetam 500mg twice a day
  Other Names: Keppra

SUMMARY:
Patients with Alzheimer's disease (AD) are increasingly recognized to have seizures in addition to cognitive decline. Seizures may contribute to memory problems as well as other symptoms common in AD like agitation, depression, or apathy. These symptoms are collectively called neuro-psychiatric symptoms. Studies of magnetic resonance imaging (MRI) in patients with AD have suggested that injury to certain parts of the brain can cause these neuro-psychiatric symptoms. Based on this evidence, the investigators hypothesize that seizures can also cause neuro-psychiatric symptoms in patients with AD and may be related to the injury seen on MRI.

The current study will follow participants for 1 year and will involve participants with AD who also have neuro-psychiatric symptoms. Participants will be examined with three brain wave studies to assess for seizure-like activity. Participants with seizure-like activity will all receive levetiracetam for 1 year. All participants will have their neuro-psychiatric symptoms, cognitive abilities, quality of life, and AD severity assessed throughout the year. The investigators plan to determine if levetiracetam changes the severity of the participants' neuro-psychiatric symptoms compared to their baseline as well as compared to participants without seizure-like activity. 65 participants will need to be recruited to test the study hypotheses. The study will take place at Walter Reed National Military Medical Center.

DETAILED DESCRIPTION:
Alzheimer's Disease (AD) has long been known to carry an increased risk of seizure, with early estimates suggesting patients with AD have a 10-22% risk at least one unprovoked seizure and an 8- to 10-fold higher seizure rate over the general population. Retrospective data has suggested that the onset of both clinical seizure and abnormal discharge on electroencephalogram (EEG) may cluster around or even precede the onset of cognitive decline. With extended EEG and/or 1-hour magnetoencephalogram (MEG), up to 42% of patients with AD have evidence of subclinical seizure or epileptiform discharges, two-thirds of which were identified only during sleep. Recent evidence has also found a much higher incidence of dyscognitive seizure (47%) and other nonconvulsive semiologies (55%) than previously reported, including jamais vu, déjà vu, sensory phenomenon, speech arrest/aphasia, and amnestic spells.

A particularly problematic aspect of dementia in general and AD in particular is neuropsychiatric symptoms. Neuropsychiatric symptoms increase with duration and severity of dementia, observed in as much as 60-90% of these patients. To some extent, neuropsychiatric symptoms may also be associated with focal dysfunction, particularly of the non-dominant fronto-temporal lobes. Seizure or transient epileptiform discharges, then, might explain some of the neuropsychiatric manifestations associated with AD, especially since the most common areas of discharge are the fronto-temporal lobes in AD. Neuropsychiatric symptoms and their causes are of particular concern in the management of patients with AD given the strain on patients and families and their high association with nursing home placement.

This study will complete up to 3 serial EEGs on each participant, and all participants with epileptiform activity identified on EEG will be started on levetiracetam. All participants will be followed with serial neuro-psychiatric symptom, cognitive, severity, and quality-of-life metrics in order to analyze the effect of levetiracetam on these measures over 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Meet the National Institute of Aging-Alzheimer's Association criteria for probable AD
* Twelve-item Neuropsychiatric Inventory with score 4 or greater
* MMSE <26
* Stable doses current medications, including acetylcholinesterase inhibitors if applicable, for at least 4 weeks prior to trial entry
* Reliable caregiver willing and available to assist with medication administration, outcome measures
* MRI completed with no evidence of potential seizure focus as outlined in the exclusion criteria

Exclusion Criteria:

* Imaging suggestive of potential seizure focus or alternative cause of dementia
* Previous Epilepsy diagnosis
* Use of anti-epileptic medication for any indication within previous three months
* History of head trauma with loss of consciousness more than 30 minutes
* Alcohol/Substance abuse within 5 years of dementia onset or previous 5 years
* History of Korsakoff's syndrome
* History of encephalitis/meningitis
* Female participant who is pregnant, lactating or planning pregnancy during trial
* Scheduled elective surgery or other procedures requiring general anesthesia during the trial
* Participant with life expectancy of less than 12 months
* Any cancer requiring current chemotherapy
* Known allergy or history of previous adverse reaction to levetiracetam
* Major depression or other significant behavioral disturbance preceding Alzheimer's Disease diagnosis
* Enrollment in another clinical treatment trial
* Laboratory evidence of an alternative cause of dementia or which might preclude treatment, including untreated vitamin B12 deficiency, untreated hypothyroidism, syphilis, positive human immunodeficiency virus testing, end-stage renal disease on dialysis, significant renal impairment (creatinine clearance <75 ml/minute), or liver function tests >2x upper limit of normal within the preceding three months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change in Neuropsychiatric Inventory Score (NPI) | Assessed at enrollment, week 7, week 15, week 27, and month 12
  Neuropsychiatric Symptom Metric

SECONDARY OUTCOMES:
Change in Clinical Dementia Rating Sum of Boxes (CDR-SOB) | Assessed at enrollment, week 7, week 15, week 27, and month 12
  Patient/Informant AD Severity Metric
Change in Alzheimer's Disease Cooperative study - Clinical Global Impression of Change (ADCS-CGIC) | Assessed at enrollment, week 7, week 15, week 27, and month 12
  Clinician AD Severity Metric
Change in EuroQol 5-Dimension (EQ-5D) | Assessed at enrollment, week 7, week 15, week 27, and month 12
  Quality of Life Metric
Change in Mini-Mental State Exam (MMSE) | Assessed at enrollment, week 7, week 15, week 27, and month 12
  Cognitive Ability Metric

CONTACTS AND LOCATIONS:
Overall Officials: Timothy R Malone, MD, Principal Investigator — Walter Reed National Military Medical Center
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hauser WA, Morris ML, Heston LL, Anderson VE. Seizures and myoclonus in patients with Alzheimer's disease. Neurology. 1986 Sep;36(9):1226-30. doi: 10.1212/wnl.36.9.1226. PMID 3092131
- [Background] Romanelli MF, Morris JC, Ashkin K, Coben LA. Advanced Alzheimer's disease is a risk factor for late-onset seizures. Arch Neurol. 1990 Aug;47(8):847-50. doi: 10.1001/archneur.1990.00530080029006. PMID 2375689
- [Background] Volicer L, Smith S, Volicer BJ. Effect of seizures on progression of dementia of the Alzheimer type. Dementia. 1995 Sep-Oct;6(5):258-63. doi: 10.1159/000106956. PMID 8528372
- [Background] Mendez M, Lim G. Seizures in elderly patients with dementia: epidemiology and management. Drugs Aging. 2003;20(11):791-803. doi: 10.2165/00002512-200320110-00001. PMID 12964886
- [Background] Amatniek JC, Hauser WA, DelCastillo-Castaneda C, Jacobs DM, Marder K, Bell K, Albert M, Brandt J, Stern Y. Incidence and predictors of seizures in patients with Alzheimer's disease. Epilepsia. 2006 May;47(5):867-72. doi: 10.1111/j.1528-1167.2006.00554.x. PMID 16686651
- [Background] Palop JJ, Mucke L. Epilepsy and cognitive impairments in Alzheimer disease. Arch Neurol. 2009 Apr;66(4):435-40. doi: 10.1001/archneurol.2009.15. Epub 2009 Feb 9. PMID 19204149
- [Background] Scarmeas N, Honig LS, Choi H, Cantero J, Brandt J, Blacker D, Albert M, Amatniek JC, Marder K, Bell K, Hauser WA, Stern Y. Seizures in Alzheimer disease: who, when, and how common? Arch Neurol. 2009 Aug;66(8):992-7. doi: 10.1001/archneurol.2009.130. PMID 19667221
- [Background] Campion D, Flaman JM, Brice A, Hannequin D, Dubois B, Martin C, Moreau V, Charbonnier F, Didierjean O, Tardieu S, et al. Mutations of the presenilin I gene in families with early-onset Alzheimer's disease. Hum Mol Genet. 1995 Dec;4(12):2373-7. doi: 10.1093/hmg/4.12.2373. PMID 8634712
- [Background] Fox NC, Kennedy AM, Harvey RJ, Lantos PL, Roques PK, Collinge J, Hardy J, Hutton M, Stevens JM, Warrington EK, Rossor MN. Clinicopathological features of familial Alzheimer's disease associated with the M139V mutation in the presenilin 1 gene. Pedigree but not mutation specific age at onset provides evidence for a further genetic factor. Brain. 1997 Mar;120 ( Pt 3):491-501. doi: 10.1093/brain/120.3.491. PMID 9126060
- [Background] Lopera F, Ardilla A, Martinez A, Madrigal L, Arango-Viana JC, Lemere CA, Arango-Lasprilla JC, Hincapie L, Arcos-Burgos M, Ossa JE, Behrens IM, Norton J, Lendon C, Goate AM, Ruiz-Linares A, Rosselli M, Kosik KS. Clinical features of early-onset Alzheimer disease in a large kindred with an E280A presenilin-1 mutation. JAMA. 1997 Mar 12;277(10):793-9. PMID 9052708
- [Background] Axelman K, Basun H, Lannfelt L. Wide range of disease onset in a family with Alzheimer disease and a His163Tyr mutation in the presenilin-1 gene. Arch Neurol. 1998 May;55(5):698-702. doi: 10.1001/archneur.55.5.698. PMID 9605727
- [Background] Janssen JC, Hall M, Fox NC, Harvey RJ, Beck J, Dickinson A, Campbell T, Collinge J, Lantos PL, Cipolotti L, Stevens JM, Rossor MN. Alzheimer's disease due to an intronic presenilin-1 (PSEN1 intron 4) mutation: A clinicopathological study. Brain. 2000 May;123 ( Pt 5):894-907. doi: 10.1093/brain/123.5.894. PMID 10775535
- [Background] Cabrejo L, Guyant-Marechal L, Laquerriere A, Vercelletto M, De la Fourniere F, Thomas-Anterion C, Verny C, Letournel F, Pasquier F, Vital A, Checler F, Frebourg T, Campion D, Hannequin D. Phenotype associated with APP duplication in five families. Brain. 2006 Nov;129(Pt 11):2966-76. doi: 10.1093/brain/awl237. Epub 2006 Sep 7. PMID 16959815
- [Background] Irizarry MC, Jin S, He F, Emond JA, Raman R, Thomas RG, Sano M, Quinn JF, Tariot PN, Galasko DR, Ishihara LS, Weil JG, Aisen PS. Incidence of new-onset seizures in mild to moderate Alzheimer disease. Arch Neurol. 2012 Mar;69(3):368-72. doi: 10.1001/archneurol.2011.830. PMID 22410444
- [Background] Mendez MF, Catanzaro P, Doss RC, ARguello R, Frey WH 2nd. Seizures in Alzheimer's disease: clinicopathologic study. J Geriatr Psychiatry Neurol. 1994 Oct-Dec;7(4):230-3. doi: 10.1177/089198879400700407. PMID 7826492
- [Background] Risse SC, Lampe TH, Bird TD, Nochlin D, Sumi SM, Keenan T, Cubberley L, Peskind E, Raskind MA. Myoclonus, seizures, and paratonia in Alzheimer disease. Alzheimer Dis Assoc Disord. 1990 Winter;4(4):217-25. doi: 10.1097/00002093-199040400-00003. PMID 2264979
- [Background] Vossel KA, Beagle AJ, Rabinovici GD, Shu H, Lee SE, Naasan G, Hegde M, Cornes SB, Henry ML, Nelson AB, Seeley WW, Geschwind MD, Gorno-Tempini ML, Shih T, Kirsch HE, Garcia PA, Miller BL, Mucke L. Seizures and epileptiform activity in the early stages of Alzheimer disease. JAMA Neurol. 2013 Sep 1;70(9):1158-66. doi: 10.1001/jamaneurol.2013.136. PMID 23835471
- [Background] Vossel KA, Ranasinghe KG, Beagle AJ, Mizuiri D, Honma SM, Dowling AF, Darwish SM, Van Berlo V, Barnes DE, Mantle M, Karydas AM, Coppola G, Roberson ED, Miller BL, Garcia PA, Kirsch HE, Mucke L, Nagarajan SS. Incidence and impact of subclinical epileptiform activity in Alzheimer's disease. Ann Neurol. 2016 Dec;80(6):858-870. doi: 10.1002/ana.24794. Epub 2016 Nov 7. PMID 27696483
- [Background] Forstl H, Burns A, Levy R, Cairns N, Luthert P, Lantos P. Neurologic signs in Alzheimer's disease. Results of a prospective clinical and neuropathologic study. Arch Neurol. 1992 Oct;49(10):1038-42. doi: 10.1001/archneur.1992.00530340054018. PMID 1417511
- [Background] Palop JJ, Chin J, Roberson ED, Wang J, Thwin MT, Bien-Ly N, Yoo J, Ho KO, Yu GQ, Kreitzer A, Finkbeiner S, Noebels JL, Mucke L. Aberrant excitatory neuronal activity and compensatory remodeling of inhibitory hippocampal circuits in mouse models of Alzheimer's disease. Neuron. 2007 Sep 6;55(5):697-711. doi: 10.1016/j.neuron.2007.07.025. PMID 17785178
- [Background] Sanchez PE, Zhu L, Verret L, Vossel KA, Orr AG, Cirrito JR, Devidze N, Ho K, Yu GQ, Palop JJ, Mucke L. Levetiracetam suppresses neuronal network dysfunction and reverses synaptic and cognitive deficits in an Alzheimer's disease model. Proc Natl Acad Sci U S A. 2012 Oct 16;109(42):E2895-903. doi: 10.1073/pnas.1121081109. Epub 2012 Aug 6. PMID 22869752
- [Background] Kleen JK, Scott RC, Holmes GL, Roberts DW, Rundle MM, Testorf M, Lenck-Santini PP, Jobst BC. Hippocampal interictal epileptiform activity disrupts cognition in humans. Neurology. 2013 Jul 2;81(1):18-24. doi: 10.1212/WNL.0b013e318297ee50. Epub 2013 May 17. PMID 23685931
- [Background] McAreavey MJ, Ballinger BR, Fenton GW. Epileptic seizures in elderly patients with dementia. Epilepsia. 1992 Jul-Aug;33(4):657-60. doi: 10.1111/j.1528-1157.1992.tb02343.x. PMID 1628580
- [Background] Heyman A, Wilkinson WE, Hurwitz BJ, Helms MJ, Haynes CS, Utley CM, Gwyther LP. Early-onset Alzheimer's disease: clinical predictors of institutionalization and death. Neurology. 1987 Jun;37(6):980-4. doi: 10.1212/wnl.37.6.980. PMID 3587649
- [Background] Oh H, Jagust WJ. Frontotemporal network connectivity during memory encoding is increased with aging and disrupted by beta-amyloid. J Neurosci. 2013 Nov 20;33(47):18425-37. doi: 10.1523/JNEUROSCI.2775-13.2013. PMID 24259567
- [Background] Huijbers W, Mormino EC, Schultz AP, Wigman S, Ward AM, Larvie M, Amariglio RE, Marshall GA, Rentz DM, Johnson KA, Sperling RA. Amyloid-beta deposition in mild cognitive impairment is associated with increased hippocampal activity, atrophy and clinical progression. Brain. 2015 Apr;138(Pt 4):1023-35. doi: 10.1093/brain/awv007. Epub 2015 Feb 11. PMID 25678559
- [Background] Scharfman HE. Alzheimer's disease and epilepsy: insight from animal models. Future Neurol. 2012 Mar 1;7(2):177-192. doi: 10.2217/fnl.12.8. PMID 22723738
- [Background] Savva GM, Zaccai J, Matthews FE, Davidson JE, McKeith I, Brayne C; Medical Research Council Cognitive Function and Ageing Study. Prevalence, correlates and course of behavioural and psychological symptoms of dementia in the population. Br J Psychiatry. 2009 Mar;194(3):212-9. doi: 10.1192/bjp.bp.108.049619. PMID 19252147
- [Background] Gitlin LN, Kales HC, Lyketsos CG. Nonpharmacologic management of behavioral symptoms in dementia. JAMA. 2012 Nov 21;308(19):2020-9. doi: 10.1001/jama.2012.36918. PMID 23168825
- [Background] Mega MS, Cummings JL, Fiorello T, Gornbein J. The spectrum of behavioral changes in Alzheimer's disease. Neurology. 1996 Jan;46(1):130-5. doi: 10.1212/wnl.46.1.130. PMID 8559361
- [Background] Lyketsos CG, Steinberg M, Tschanz JT, Norton MC, Steffens DC, Breitner JC. Mental and behavioral disturbances in dementia: findings from the Cache County Study on Memory in Aging. Am J Psychiatry. 2000 May;157(5):708-14. doi: 10.1176/appi.ajp.157.5.708. PMID 10784462
- [Background] Lyketsos CG, Lopez O, Jones B, Fitzpatrick AL, Breitner J, DeKosky S. Prevalence of neuropsychiatric symptoms in dementia and mild cognitive impairment: results from the cardiovascular health study. JAMA. 2002 Sep 25;288(12):1475-83. doi: 10.1001/jama.288.12.1475. PMID 12243634
- [Background] Sink KM, Covinsky KE, Newcomer R, Yaffe K. Ethnic differences in the prevalence and pattern of dementia-related behaviors. J Am Geriatr Soc. 2004 Aug;52(8):1277-83. doi: 10.1111/j.1532-5415.2004.52356.x. PMID 15271114
- [Background] Peters KR, Rockwood K, Black SE, Bouchard R, Gauthier S, Hogan D, Kertesz A, Loy-English I, Beattie BL, Sadovnick AD, Feldman HH. Characterizing neuropsychiatric symptoms in subjects referred to dementia clinics. Neurology. 2006 Feb 28;66(4):523-8. doi: 10.1212/01.wnl.0000198255.84842.06. PMID 16505306
- [Background] Rosen HJ, Allison SC, Schauer GF, Gorno-Tempini ML, Weiner MW, Miller BL. Neuroanatomical correlates of behavioural disorders in dementia. Brain. 2005 Nov;128(Pt 11):2612-25. doi: 10.1093/brain/awh628. Epub 2005 Sep 29. PMID 16195246
- [Background] Gallagher-Thompson D, Brooks JO 3rd, Bliwise D, Leader J, Yesavage JA. The relations among caregiver stress, "sundowning" symptoms, and cognitive decline in Alzheimer's disease. J Am Geriatr Soc. 1992 Aug;40(8):807-10. doi: 10.1111/j.1532-5415.1992.tb01853.x. PMID 1634724
- [Background] Scarmeas N, Brandt J, Blacker D, Albert M, Hadjigeorgiou G, Dubois B, Devanand D, Honig L, Stern Y. Disruptive behavior as a predictor in Alzheimer disease. Arch Neurol. 2007 Dec;64(12):1755-61. doi: 10.1001/archneur.64.12.1755. PMID 18071039
- [Background] O'Donnell BF, Drachman DA, Barnes HJ, Peterson KE, Swearer JM, Lew RA. Incontinence and troublesome behaviors predict institutionalization in dementia. J Geriatr Psychiatry Neurol. 1992 Jan-Mar;5(1):45-52. doi: 10.1177/002383099200500108. PMID 1571074
- [Background] Morriss RK, Rovner BW, Folstein MF, German PS. Delusions in newly admitted residents of nursing homes. Am J Psychiatry. 1990 Mar;147(3):299-302. doi: 10.1176/ajp.147.3.299. PMID 2309945
- [Background] Scarmeas N, Brandt J, Albert M, Hadjigeorgiou G, Papadimitriou A, Dubois B, Sarazin M, Devanand D, Honig L, Marder K, Bell K, Wegesin D, Blacker D, Stern Y. Delusions and hallucinations are associated with worse outcome in Alzheimer disease. Arch Neurol. 2005 Oct;62(10):1601-8. doi: 10.1001/archneur.62.10.1601. PMID 16216946
- [Background] McKhann GM, Knopman DS, Chertkow H, Hyman BT, Jack CR Jr, Kawas CH, Klunk WE, Koroshetz WJ, Manly JJ, Mayeux R, Mohs RC, Morris JC, Rossor MN, Scheltens P, Carrillo MC, Thies B, Weintraub S, Phelps CH. The diagnosis of dementia due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):263-9. doi: 10.1016/j.jalz.2011.03.005. Epub 2011 Apr 21. PMID 21514250
- [Background] Ponomareva NV, Korovaitseva GI, Rogaev EI. EEG alterations in non-demented individuals related to apolipoprotein E genotype and to risk of Alzheimer disease. Neurobiol Aging. 2008 Jun;29(6):819-27. doi: 10.1016/j.neurobiolaging.2006.12.019. Epub 2007 Feb 12. PMID 17293007
- [Background] Gorno-Tempini ML, Hillis AE, Weintraub S, Kertesz A, Mendez M, Cappa SF, Ogar JM, Rohrer JD, Black S, Boeve BF, Manes F, Dronkers NF, Vandenberghe R, Rascovsky K, Patterson K, Miller BL, Knopman DS, Hodges JR, Mesulam MM, Grossman M. Classification of primary progressive aphasia and its variants. Neurology. 2011 Mar 15;76(11):1006-14. doi: 10.1212/WNL.0b013e31821103e6. Epub 2011 Feb 16. PMID 21325651
- [Background] Mendez MF, Ghajarania M, Perryman KM. Posterior cortical atrophy: clinical characteristics and differences compared to Alzheimer's disease. Dement Geriatr Cogn Disord. 2002;14(1):33-40. doi: 10.1159/000058331. PMID 12053130
- [Background] Wessels AM, Siemers ER, Yu P, Andersen SW, Holdridge KC, Sims JR, Sundell K, Stern Y, Rentz DM, Dubois B, Jones RW, Cummings J, Aisen PS. A Combined Measure of Cognition and Function for Clinical Trials: The Integrated Alzheimer's Disease Rating Scale (iADRS). J Prev Alzheimers Dis. 2015 Dec 1;2(4):227-241. doi: 10.14283/jpad.2015.82. PMID 27019841